CLINICAL TRIAL: NCT05564507
Title: A Multicenter Randomized Study to Assess the Impact of SIMULation-bAsed Training on Transoesophageal echocardiOgraphy leaRning for Cardiology Fellows
Brief Title: Effectiveness of Simulation-based Training on Transoesophageal Echocardiography Learning
Acronym: SIMULATOR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Groupe des jeunes de la filiale d'imagerie cardiovasculaire (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: JFIC001
Record Dates: First submitted 2022-08-31; First posted 2022-10-03 (Actual); Last update posted 2022-10-03 (Actual); Status verified 2022-09

CONDITIONS: Knowledge, Attitudes, Practice; Cardiovascular Diseases; Valvular Heart Disease
Keywords: Simulation-based training; Education; Transesophageal echocardiography; Simulation
MeSH Terms: conditions — Behavior; Cardiovascular Diseases; Heart Valve Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TEE simulation-based training group (Experimental): All participants of the TEE simulation group received:
  1) a traditional didactic training using e-learning with a national free-access online course; and 2) two teaching sessions using a TEE simulator for 2 hours per session.
  Interventions: Diagnostic Test: TEE simulation-based training
- TEE traditional group (No Intervention): All participants of the TEE traditional group received only a traditional didactic training using e-learning with a national free-access online course (same e-learning program allocated for the TEE simulation group).

INTERVENTIONS:
Diagnostic Test: TEE simulation-based training — All participants of the TEE simulation-based training group received:
  1. a traditional didactic training using e-learning with a national free-access online course;
  2. two teaching sessions using a TEE simulator for 2 hours per session. The simulation session will involve standardized initial teaching of normal cardiac, including anatomy of mitral valve with some mitral regurgitation cases, aortic valve, tricuspid valve, interatrial septum, and left atrial appendage, and demonstration of image acquisition by the teacher (time duration: 30 min). The duration of each session was 2 h with a 6:1 student to instructor ratio. Each subject had a dedicated 20 min of hands-on to manipulate the probe and undertake a sequential TEE examination under the supervision of the teacher. Other participants could watch their colleagues working on the TEE simulator.
  Arms: TEE simulation-based training group

SUMMARY:
Background:

Simulation-based training in transesophageal echocardiography (TEE) seems promising. However, data are limited to non-randomized or single-center studies.

Objectives:

This large multicenter randomized, parallel-group, unblinded, study will assess the impact of simulation-based versus traditional teaching on TEE knowledge and performance for medical fellows in cardiology.

Eligibility:

* All consecutive fellows in cardiology of all training levels (year 1-4)
* who have never performed a TEE alone

Design:

* Multicenter, parallel-group, unblinded, randomized study with a prospective enrollment of all consecutive fellows in cardiology of all training level (year 1 to 4) who were recruited in 42 centers throughout France.
* Randomization with stratification by center will be performed at the individual (fellow) level in 1:1 ratio to assign all the fellows to the traditional group or to the TEE simulation-based training group.
* Each participant will complete two different tests during the study: 1) a pre-training test before starting the educational program; and 2) a final test performed 3 months after the end of the educational program. Each of these tests will include a theoretical test and a practical test on a TEE simulator.
* The coprimary outcomes of the study to compare the two groups will be the scores in the final theoretical and practical tests after the training will be completed.

DETAILED DESCRIPTION:
Background:

Recent studies suggested that simulation-based transesophageal echocardiography (TEE) teaching is displaying significant benefit over conventional methods based on academic lectures in terms of improving TEE skills and accelerating learning. However, evidence on the impact of simulation-based training in TEE is scarce. Indeed, all the studies assessing the effectiveness of TEE simulation-based teaching were non-randomized or randomized with limited single-center sample size

Objectives:

This large multicenter randomized, parallel-group, unblinded, study will assess the impact of simulation-based versus traditional teaching on TEE knowledge and performance for medical fellows in cardiology.

Methods:

The SIMULATOR study will be a multicenter, parallel-group, unblinded, randomized study including all consecutive fellows in cardiology of all training level (year 1 to 4) who will be randomized (1:1) to either a TEE simulation group or to a traditional group through 42 French centers. Fellows who had already performed a TEE alone, with or without supervision, will be excluded. All the fellows will give their consent to participate to the study and agree to provide their honest answers and thoughts about their skills and confidence about their practices.

Each participant will complete two different tests during the study: 1) a pre-training test before starting the educational program; and 2) a final test performed 3 months after the end of the educational program. Each of these tests will include a theoretical test and a practical test on a TEE simulator.

Endpoints:

The coprimary endpoints of the study will be the difference in the final theoretical and practical tests score after the training between the two groups. The secondary endpoints will be the difference in change in theoretical and practical tests scores from pre- to final training. In addition, we will assess the global score defined as the sum of the theoretical test and the practical test scores, the TEE exam duration, and the self-assessment of proficiency of the fellows.

Sample size calculation:

Details regarding the determination of the sample size have been reported previously. Based on recent available literature and considering normalized 0-100 points score ranges for the two co-primary outcomes, a minimally important difference of 5 points (standard deviation 7 points) will be considered for the difference in change from pre- to post-training scores in theoretical and practical tests between the two randomized groups. Under these assumptions, a sample size of 50 subjects per group (for an overall population of 100 participants) will provide 90% power to detect a statistically significant difference between the two groups at a significance level of alpha = 2.5%, applying a Bonferroni correction to account for multiple testing of the two co-primary outcomes.

ELIGIBILITY:
Inclusion Criteria:

* All consecutive fellows in cardiology of all training levels (year 1-4) who have never performed a TEE alone.

Exclusion Criteria:

* Fellows who had already performed a TEE alone, with or without supervision, were excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 385 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-02-01 (Actual)

PRIMARY OUTCOMES:
Difference in the final theoretical test score after the training between the two groups. | 3 months after completion of the training program
  Each resident completed two sets of tests during the study:
  1) a pre-training test before starting the training program to assess the baseline TEE level of each resident; and 2) a final test performed 3 months after the end of the training program.
  The theoretical test included 20 video-based questions online that evaluate recognition of standard TEE views, normal anatomy and some pathological cases as already described. The fellows were given 90 seconds for each question to choose the best answer out of a multiple-choice of 5 propositions. Each question was scored on 5 points (5 points if all the propositions were correct and 0 point if at least one error was observed), for a total of 100 points per test.
Difference in the final practical test score after the training between the two groups. | 3 months after completion of the training program
  Each resident completed two sets of tests during the study:
  1) a pre-training test before starting the training program to assess the baseline TEE level of each resident; and 2) a final test performed 3 months after the end of the training program. Each of these tests included a practical test on a TEE simulator .
  Immediately after each theoretical test (pre-training and final tests), all fellows underwent the practical test. The fellows were asked to show ten basic views on a TEE simulator, as previously described, and were given a maximum of one minute for each view. The practical test was stopped after a maximum of 10 minutes. Each view was scored on 10 points using the modified Ferrero grading scale, for a total of 100 points per practical test.

SECONDARY OUTCOMES:
Difference in change in theoretical test scores from pre- to final training | 3 months after completion of the training program
  Difference in change in theoretical test scores from pre- to final training.
  The theoretical test included 20 video-based questions online that evaluate recognition of standard TEE views, normal anatomy and some pathological cases as already described. The fellows were given 90 seconds for each question to choose the best answer out of a multiple-choice of 5 propositions. Each question was scored on 5 points (5 points if all the propositions were correct and 0 point if at least one error was observed), for a total of 100 points per test.
Difference in change in practical test scores from pre- to final training | 3 months after completion of the training program
  Difference in change in practical test scores from pre- to final training.
  To standardize the training and the practical test on TEE simulator, all trainers followed a dedicated webinar of 30 minutes presenting the entire content of each session and the final test. Immediately after each theoretical test (pre-training and final tests), all fellows underwent the practical test. The fellows were asked to show ten basic views on a TEE simulator, as previously described, and were given a maximum of one minute for each view. The teacher timed the duration between the TEE probe introduction and obtention by the trainee of all ten views required. The practical test was stopped after a maximum of 10 minutes. Each view was scored on 10 points using the modified Ferrero grading scale, for a total of 100 points per practical test.
Difference in the final global score after the training between the two groups. | 3 months after completion of the training program
  The global score was defined as the sum of the theoretical test and the practical test scores, the TEE exam duration, and the self-assessment of proficiency of the fellows.
Difference in TEE exam duration after the training between the two groups. | 3 months after completion of the training program
  The trainer measured the TEE exam duration during the practical test using simulator.
Self-assessment of proficiency of the fellows | 3 months after completion of the training program
  The self-assessment of proficiency of all the fellows was assessed with four standardised questions asked before and immediately after the training program:
  1. "Do you feel ready to perform a TEE alone?",
  2. "Do you feel confident to perform a TEE alone?",
  3. "Do you feel comfortable with TEE probe introduction?" and 4) "Do you feel comfortable with TEE probe manipulation?". Each question was graded from 1 (lower grade) to 5 (higher grade).
  In the simulation group, satisfaction after the simulation training was assessed by an anonymous questionnaire including six statements on different aspects of the training, as already published.

CONTACTS AND LOCATIONS:
Locations (1):
- Augustin Coisne, Lille, Hauts-de-France, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pezel T, Dreyfus J, Mouhat B, Thebaut C, Audureau E, Bernard A, Badie YL, Bohbot Y, Fard D, Nguyen LS, Monteil C, Biere L, Le Ven F, Canu M, Ribeyrolles S, Mion B, Bazire B, Fauvel C, Cautela J, Cambet T, Le Tourneau T, Donal E, Lafitte S, Magne J, Mansencal N, Coisne A; SIMULATOR investigators. Effectiveness of Simulation-Based Training on Transesophageal Echocardiography Learning: The SIMULATOR Randomized Clinical Trial. JAMA Cardiol. 2023 Mar 1;8(3):248-256. doi: 10.1001/jamacardio.2022.5016. PMID 37070491